CLINICAL TRIAL: NCT00258583
Title: Dorothy P. and Richard P Simmons Center for Interstitial Lung Disease Research Registry
Brief Title: Dorothy P. and Richard P. Simmons Center for ILD Research Registry
Acronym: ILDRR
Status: Recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Kevin F. Gibson, Professor of Medicine, University of Pittsburgh
Other Study IDs: STUDY20030050
Record Dates: First submitted 2005-11-23; First posted 2005-11-24 (Estimated); Last update posted 2025-10-29 (Actual); Status verified 2025-09

CONDITIONS: Lung Diseases, Interstitial
Keywords: "Lung[A04.400]"
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to place past, current, and future medical record information into the UPMC Simmons Center for Interstitial Lung Disease Research Registry.

DETAILED DESCRIPTION:
This study gives participant's permission to allow the staff at the Dorothy P. and Richard P. Simmons Center for Interstitial Lung Disease to to place past, current, and future medical record information into a UPMC Simmons Center for Interstitial Lung Disease Research Registry. By placing the medical record information of many patients into a research registry, researchers will be able to conduct research studies directed at increasing our knowledge about interstitial lung disease. It is anticipated that the research registry will assist out investigators by allowing researchers to review and study the medical records of many individuals to answer questions about interstitial lung disease and its treatment. In addition, it will help researchers identify and recruit patients for participation in future research studies.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who are seeking treatment at the UPMC Simmons Center for Interstitial Lung Disease
* 18 years of age or older

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population can be described as any adult being seen by a physician at the Simmons Center for interstitial lung disease who has been diagnosed with an Interstitial Lung Disease.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2003-10; Primary Completion 2035-07 (Estimated); Study Completion 2035-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin F Gibson, MD, Principal Investigator — University of Pittsburgh - UPMC Simmons Center for Interstitial Lung Disease
Locations (1):
- Michelle F MacPherson, Pittsburgh, Pennsylvania, United States

REFERENCES:
- See also: The Dorothy P. and Richard P. Simmons Center for Interstitial Lung Disease is designed to provide patient-friendly advice and support for people with idiopathic pulmonary fibrosis. — http://www.upmc.com/services/pulmonology/interstitial-lung-disease/